CLINICAL TRIAL: NCT00465257
Title: Efficacy of Artesunate + Amodiaquine Four Years After Its Introduction as New Treatment Policy for Uncomplicated Plasmodium Falciparum Malaria in Zanzibar
Brief Title: Efficacy of Artesunate + Amodiaquine Four Years After Its Introduction in Zanzibar
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to lack of malaria patients in Zanzibar the study has been suspended.
Sponsor: Karolinska University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: ACOIII
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination

INTERVENTIONS:
Drug: artesunate + amodiaquine

SUMMARY:
The purpose of this study is to assess the efficacy of artesuante + amodiaquine four years after its introduction as first line treatment for uncomplicated childhood malaria in Zanzibar. The hypothesis is that the treatment has a polymerase chain reaction (PCR)adjusted parasitological cure rate of at least 85% 42 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age below 60 months
* Weight ≥5kg
* No general danger signs or severe malaria present (see 4.4.2.1 & 4.4.2.2)
* History of fever within 24 hours OR axillary temperature ≥ 37.5Cº
* No other cause of fever is detectable
* No severe malnutrition
* Presence of P. falciparum asexual parasite density between 2000- 200,000/ul
* Guardian/Patient has understood the procedures of the study and is willing to participate
* Patient able to come for stipulated follow up visits and has easy access to the Study Site

Exclusion Criteria:

* Not able to drink or breastfeed
* Persistent Vomiting
* Recent history of convulsions
* Lethargic or unconscious
* Unable to sit or stand (as appropriate for age)
* History of allergy to test drugs
* History of intake of any drugs other than paracetamol and aspirin within 3 days

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2007-05

PRIMARY OUTCOMES:
PCR adjusted parasitological cure rate by day 42.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Björkman, Professor, Study Director — Karolinska UH; Guida Rotlland, MD, MPH, Principal Investigator — Karolinska UH
Locations (1):
- Kivunge Cottage Hospital, Kivunge, North A District, Zanzibar, Tanzania